CLINICAL TRIAL: NCT05974670
Title: Early Warning Value of Consumer Wearable Devices in Chronic Obstructive Pulmonary Disease Exacerbation: An Evaluation Study
Brief Title: Early Warning Value of Consumer Wearable Devices in AECOPD
Acronym: EWVCWDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021397-20220703
Record Dates: First submitted 2022-09-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: COPD
Keywords: COPD; AECOPD; Consumer wearable device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wearing device: The subjects are required to fill in the COPD symptom diary every day, and conducted online or offline follow-up at the 4th, 8th, 12th, 16th, 20th, and 24th weeks after enrollment. The physiological parameters of wearable devices, including pulse rate, blood oxygen saturation, physical activity, electrocardiogram, and sleep, will be continuously collected during the study.
  Interventions: Device: Consumer wearable device

INTERVENTIONS:
Device: Consumer wearable device — The subjects are required to wear the consumer wearable devices continuously during the whole study period. The device can provided several physiological parameters, including pulse rate, blood oxygen saturation, physical activity, electrocardiogram, and sleep.

SUMMARY:
This is a prospective, multi-center cohort study. 150 subjects with COPD and in stable stage will be included. Wearable device's physiological parameters will be continually collected, the investigators aim to explore whether consumer wearable devices are useful for early warning deterioration of COPD.

DETAILED DESCRIPTION:
This is a prospective cohort study. 150 subjects aged 35～80y with stable COPD will be recruited. After enrollment, subjects wear consumer wearable devices and install APP on their mobile phones. The first 7 days of wearing are to evaluate the stability of data collection and the subject compliance, and to correct the wrong wearing. The subjects are required to fill in the COPD symptom diary every day, and conducted online or offline follow-up at the 4th, 8th, 12th, 16th, 20th, and 24th weeks after enrollment. The physiological parameters of wearable devices, including pulse rate, blood oxygen saturation, physical activity, electrocardiogram, and sleep, will be continuously collected during the study. The Department of Respiratory and Critical Care of Peking University First Hospital is responsible for this research. Primary outcome is the moderate or more severe COPD acute exacerbation events. The purpose of this study is to use consumer wearable devices to monitor the changes of COPD, and to establish a physiological parameters model of wearable device that can predict the acute exacerbation of COPD.

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB) (2021-397). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stable COPD (refer to 2021 GOLD guidelines);
* Age between 35 and 80 years (both 35 and 80), either gender;
* A post-bronchodilator forced expiratory volume in 1 second percentage (FEV1%) predicted between 25%~80%;
* Having mobile phone which can install APP of wearable device;
* Able to engage in daily activities;

Exclusion Criteria:

* History of asthma, lung cancer, active pulmonary tuberculosis, bronchiectasis, diffuse lung disease (interstitial pneumonia, pulmonary sarcoidosis, occupational lung disease, sarcoidosis et al) and pleural disease;
* History of lobectomy and/or lung transplantation;
* Predicted life expectancy less than 3 years;
* History of serious underlying diseases (including severe psychiatric illnesses, mental disorders, neurological disorders, malignant tumors, chronic liver disease, heart failure, autoimmune diseases, chronic kidney disease);
* Alcoholism, drug or toxic solvents abuse;
* Moderate to severe anemia;
* Smoking or quitting smoking for less than 6 weeks;
* Skin pigmentation, deformity, arterial stenosis or occlusion of both upper limbs;
* Skin allergy to metal/plastic;
* Those who are participating in other clinical trials, cannot be followed up for a long time or have poor compliance.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients and inpatients from Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Moderate or more severe COPD exacerbation | 6 months
  Mild exacerbation: exacerbation requiring short-acting bronchodilator (SABD) therapy alone Moderate exacerbation: exacerbation requiring SABD and antimicrobials with or without oral corticosteroids Severe exacerbation: exacerbation requiring hospitalization or emergency, intensive care unit (ICU) treatment.

SECONDARY OUTCOMES:
Changes in symptoms (assessed by COPD Assessment Test, CAT) | 6 months
  The change in CAT score is calculated by the difference in CAT score during follow-up.
Changes in symptoms (assessed by the modified Medical Research Council (mMRC) dyspnea scores) | 6 months
  The change in mMRC score is calculated by the difference in CAT score during follow-up.
Changes in post-bronchodilator FEV1 | 6 months
  Post-bronchodilator FEV1 is measured by trained staff. The change in post-bronchodilator FEV1 is defined as the difference in FEV1 between week 24 follow-up and enrollment.
Changes in post-bronchodilator FEV1% | 6 months
  Post-bronchodilator FEV1% is measured by trained staff. The change in post-bronchodilator FEV1% is defined as the difference in FEV1 between week 24 follow-up and enrollment.
Changes in post-bronchodilator FVC | 6 months
  Post-bronchodilator FVC is measured by trained staff. The change in post-bronchodilator FVC is defined as the difference in FEV1 between week 24 follow-up and enrollment.
Changes in post-bronchodilator FVC% | 6 months
  Post-bronchodilator FVC% is measured by trained staff. The change in post-bronchodilator FVC% is defined as the difference in FEV1 between week 24 follow-up and enrollment.
Changes in post-bronchodilator FEV1/FVC | 6 months
  Post-bronchodilator FEV1/FVC is measured by trained staff. The change in post-bronchodilator FEV1/FVC is defined as the difference in FEV1 between week 24 follow-up and enrollment.
Herat rate parameters | 6 months
  A wearable device worn by the subject continuously monitors heart rate parameters, from which parameters such as heart rate can be obtained.
Blood oxygen saturation | 6 months
  A wearable device worn by the subject continuously monitors blood oxygen saturation.
Physical parameters from wearable device | 6 months
  A wearable device worn by the subject continuously monitors physical parameters, from which parameters such as steps can be obtained.
Sleep parameters from wearable device | 6 months
  A wearable device worn by the subject continuously monitors sleep parameters, from which parameters such as sleep duration can be obtained.
Wearing compliance | 6 months
  Compliance is defined as the ratio of the time of wearing a device to the total study time.
Data loss rate | 6 months
  Data loss rate

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Wang, MD., Study Chair — Peking University First Hospital
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Aerospace 731 Hospital, Beijing, Beijing Municipality
  - Beijing Miyun Hospital, Beijing, Beijing Municipality
  - Civil Aviation General Hospital, Beijing, Beijing Municipality
  - People's Hospital of Beijing Daxing District, Beijing, Beijing Municipality
  - Shichahai Community Health Service Center, Beijing, Beijing Municipality
  - The Hospital of Shunyi District Beijing, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No